CLINICAL TRIAL: NCT02719665
Title: THE OMEGA-SPM-DOSE and OMEGA-SPM-PAD: Specialized Pro-Resolving Mediators in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15-17371
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Arterial Disease; Claudication; Claudication, Intermittent; Vascular Occlusion; Vascular Calcification; Vascular Diseases; Osteoarthritis
Keywords: peripheral arterial disease; claudication; PAD; Vascular Disease; Vascular Occlusion; Vacular Calcification; intermittent claudication; Osteoarthritis
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Vascular Calcification; Vascular Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1a (OMEGA-SPM-DOSE) (Experimental): PAD patients and healthy volunteers in study for SPM Emulsion, dose-modality.
  Interventions: Dietary Supplement: SPM Emulsion, Dose-modality
- SPM - Phase 1b (OMEGA-SPM-DOSE) (Active Comparator): PAD and Osteoarthritis (OA) patients using softgel, dose-modality.
  Interventions: Dietary Supplement: SPM Softgel, Dose-Modality
- Placebo - Phase 1b (OMEGA-SPM-PLACEBO) (Placebo Comparator): PAD and Osteoarthritis (OA) patients using softgel, dose-modality.
  Interventions: Dietary Supplement: Placebo Softgel

INTERVENTIONS:
Dietary Supplement: SPM Emulsion, Dose-modality — Phase 1a Dose-Finding oral SPM administration of increasing dose (15ml, 30ml, and 60ml) by the following schedule:
  Days 1 to 5: 15 ml; Days 6 to 14: Washout, no SPM administration; Days 15 to 19: 30 ml; Days 20-28: Washout, no SPM administration; Days 29-33: 60 ml
  Other Names: Omega SPM; Specialized Pro-resolving Lipid Mediator Emulsion
  Arms: Phase 1a (OMEGA-SPM-DOSE)
Dietary Supplement: SPM Softgel, Dose-Modality — Phase 1b Dose-Finding oral softtel SPM administration of two different doses (2 softgel vs 4 softgel) Days 0 to 5: 2 SPM softgel; Days 6 to 21: Washout, no SPM administration; Days 22 to 26: 4 SPM softgel; Days 27-42: Washout, no SPM administration
  Other Names: Omega SPM Bridging
  Arms: SPM - Phase 1b (OMEGA-SPM-DOSE)
Dietary Supplement: Placebo Softgel — Days 43-47: 4 Placebo softgel; Day 48-64 Washout
  Other Names: Omega SPM Bridging
  Arms: Placebo - Phase 1b (OMEGA-SPM-PLACEBO)

SUMMARY:
The purpose of this study is to understand the effects of fish oil supplement (containing parts of omega-3 fatty acids) on inflammation. The investigators are aiming to identify which dose of the fish oil supplement is the most effective. The name of the fish oil supplement is "SPM Emulsion."

DETAILED DESCRIPTION:
The OMEGA-SPM-DOSE trial and the OMEGA-SPM-PAD trial are two parts of a pilot study which aims to investigate the effect of a novel formulation of a nutritional supplement containing highly concentrated n-3 PUFA metabolites (SPM Emulsion) on the metabolo-lipidomic profile of healthy volunteers and patients with Peripheral Arterial Disease(PAD). Ten healthy volunteers and ten patients with PAD will participate in Part 1a, the "OMEGA-SPM-DOSE Study". A follow-up, placebo controlled, prospective study on the best dosing modality determined in Phase 1a will then take place in a PAD and OA population (n=12), Phase 1b - the "OMEGA-SPM-PAD Study". Specific measurements will include targeted metabolo-lipidomic profiling, established markers of inflammation, and functional monocyte and macrophage assays. The proposed studies have the potential to provide important new insights on the role of nutritional interventions in PAD.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

-Age 20-80

PAD Patients:

* Mild claudication to rest pain (Rutherford 1-4)
* Resting or exercise ABI < 0.9 or TBI < 0.6
* Age 40 and more

OA Patients:

-Lower extremity (hip or knee) OA

Exclusion Criteria:

PAD, OA Patients and Healthy Volunteers:

* Plan to undergo surgical procedure or PVI for treatment of PAD within one month
* Evidence of active infection
* Hypersensitivity or allergy to fish or seafood
* Already on n-3 PUFA or equivalent
* Chronic liver disease, end-stage renal disease (CKD 5), or chronic inflammatory disorders
* Poorly controlled diabetes (HbA1C > 8%)
* BMI < 20 or >35
* Recent other major surgery or illness within 30 days
* Use of immunosuppressive medications or steroids
* History of organ transplantation
* Pregnancy, or plans to become pregnant, or lactating

Healthy Volunteers:

* hsCRP > 2mg/L
* Regular aspirin use
* Regular non-steroidal anti-inflammatory drug use

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Optimal Phase 1b Dose | Baseline, Day 33
  The smallest dose administered in Phase 1a participants which results in an increase in Resolution Index at least 3 times that of baseline, or the subsequent larger dose resulting in a Resolution Index greater than 2 times that of the preceding does with no increase in side effects at the larger dose.
Change in the Resolution Index | Baseline, Day 5
  Integrated metabolo-lipidomics assessment of SPM pathways: Average concentration of 15-HEPE, 18-HEPE, 4-HDHA, and 17-HDHA in plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Conte, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Grenon SM, Owens CD, Nosova EV, Hughes-Fulford M, Alley HF, Chong K, Perez S, Yen PK, Boscardin J, Hellmann J, Spite M, Conte MS. Short-Term, High-Dose Fish Oil Supplementation Increases the Production of Omega-3 Fatty Acid-Derived Mediators in Patients With Peripheral Artery Disease (the OMEGA-PAD I Trial). J Am Heart Assoc. 2015 Aug 21;4(8):e002034. doi: 10.1161/JAHA.115.002034. PMID 26296857
- [Background] Grenon SM, Owens CD, Alley H, Chong K, Yen PK, Harris W, Hughes-Fulford M, Conte MS. n-3 Polyunsaturated fatty acids supplementation in peripheral artery disease: the OMEGA-PAD trial. Vasc Med. 2013 Oct;18(5):263-74. doi: 10.1177/1358863X13503695. Epub 2013 Sep 19. PMID 24052491
- [Background] Akagi D, Chen M, Toy R, Chatterjee A, Conte MS. Systemic delivery of proresolving lipid mediators resolvin D2 and maresin 1 attenuates intimal hyperplasia in mice. FASEB J. 2015 Jun;29(6):2504-13. doi: 10.1096/fj.14-265363. Epub 2015 Mar 16. PMID 25777995
- [Background] Chatterjee A, Sharma A, Chen M, Toy R, Mottola G, Conte MS. The pro-resolving lipid mediator maresin 1 (MaR1) attenuates inflammatory signaling pathways in vascular smooth muscle and endothelial cells. PLoS One. 2014 Nov 19;9(11):e113480. doi: 10.1371/journal.pone.0113480. eCollection 2014. PMID 25409514
- [Background] Miyahara T, Runge S, Chatterjee A, Chen M, Mottola G, Fitzgerald JM, Serhan CN, Conte MS. D-series resolvin attenuates vascular smooth muscle cell activation and neointimal hyperplasia following vascular injury. FASEB J. 2013 Jun;27(6):2220-32. doi: 10.1096/fj.12-225615. Epub 2013 Feb 13. PMID 23407709
- [Background] Hudert CA, Weylandt KH, Lu Y, Wang J, Hong S, Dignass A, Serhan CN, Kang JX. Transgenic mice rich in endogenous omega-3 fatty acids are protected from colitis. Proc Natl Acad Sci U S A. 2006 Jul 25;103(30):11276-81. doi: 10.1073/pnas.0601280103. Epub 2006 Jul 17. PMID 16847262
- [Background] Recchiuti A, Codagnone M, Pierdomenico AM, Rossi C, Mari VC, Cianci E, Simiele F, Gatta V, Romano M. Immunoresolving actions of oral resolvin D1 include selective regulation of the transcription machinery in resolution-phase mouse macrophages. FASEB J. 2014 Jul;28(7):3090-102. doi: 10.1096/fj.13-248393. Epub 2014 Apr 1. PMID 24692596
- [Background] Wang X, Hjorth E, Vedin I, Eriksdotter M, Freund-Levi Y, Wahlund LO, Cederholm T, Palmblad J, Schultzberg M. Effects of n-3 FA supplementation on the release of proresolving lipid mediators by blood mononuclear cells: the OmegAD study. J Lipid Res. 2015 Mar;56(3):674-681. doi: 10.1194/jlr.P055418. Epub 2015 Jan 23. PMID 25616438
- [Background] Chiang N, Fredman G, Backhed F, Oh SF, Vickery T, Schmidt BA, Serhan CN. Infection regulates pro-resolving mediators that lower antibiotic requirements. Nature. 2012 Apr 25;484(7395):524-8. doi: 10.1038/nature11042. PMID 22538616
- [Background] Mizwicki MT, Liu G, Fiala M, Magpantay L, Sayre J, Siani A, Mahanian M, Weitzman R, Hayden EY, Rosenthal MJ, Nemere I, Ringman J, Teplow DB. 1alpha,25-dihydroxyvitamin D3 and resolvin D1 retune the balance between amyloid-beta phagocytosis and inflammation in Alzheimer's disease patients. J Alzheimers Dis. 2013;34(1):155-70. doi: 10.3233/JAD-121735. PMID 23186989
- [Background] Oh SF, Pillai PS, Recchiuti A, Yang R, Serhan CN. Pro-resolving actions and stereoselective biosynthesis of 18S E-series resolvins in human leukocytes and murine inflammation. J Clin Invest. 2011 Feb;121(2):569-81. doi: 10.1172/JCI42545. Epub 2011 Jan 4. PMID 21206090
- [Background] Serhan CN, Yang R, Martinod K, Kasuga K, Pillai PS, Porter TF, Oh SF, Spite M. Maresins: novel macrophage mediators with potent antiinflammatory and proresolving actions. J Exp Med. 2009 Jan 16;206(1):15-23. doi: 10.1084/jem.20081880. Epub 2008 Dec 22. PMID 19103881
- [Background] Serhan CN. Resolution phase of inflammation: novel endogenous anti-inflammatory and proresolving lipid mediators and pathways. Annu Rev Immunol. 2007;25:101-37. doi: 10.1146/annurev.immunol.25.022106.141647. PMID 17090225
- [Background] Serhan CN. Pro-resolving lipid mediators are leads for resolution physiology. Nature. 2014 Jun 5;510(7503):92-101. doi: 10.1038/nature13479. PMID 24899309
- [Background] Ross R. Atherosclerosis--an inflammatory disease. N Engl J Med. 1999 Jan 14;340(2):115-26. doi: 10.1056/NEJM199901143400207. No abstract available. PMID 9887164
- [Background] Tzoulaki I, Murray GD, Lee AJ, Rumley A, Lowe GD, Fowkes FG. C-reactive protein, interleukin-6, and soluble adhesion molecules as predictors of progressive peripheral atherosclerosis in the general population: Edinburgh Artery Study. Circulation. 2005 Aug 16;112(7):976-83. doi: 10.1161/CIRCULATIONAHA.104.513085. Epub 2005 Aug 8. PMID 16087797
- [Background] Beckman JA, Preis O, Ridker PM, Gerhard-Herman M. Comparison of usefulness of inflammatory markers in patients with versus without peripheral arterial disease in predicting adverse cardiovascular outcomes (myocardial infarction, stroke, and death). Am J Cardiol. 2005 Nov 15;96(10):1374-8. doi: 10.1016/j.amjcard.2005.07.041. Epub 2005 Sep 27. PMID 16275181
- [Background] Ridker PM, Stampfer MJ, Rifai N. Novel risk factors for systemic atherosclerosis: a comparison of C-reactive protein, fibrinogen, homocysteine, lipoprotein(a), and standard cholesterol screening as predictors of peripheral arterial disease. JAMA. 2001 May 16;285(19):2481-5. doi: 10.1001/jama.285.19.2481. PMID 11368701
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Plasma concentration of C-reactive protein and risk of developing peripheral vascular disease. Circulation. 1998 Feb 10;97(5):425-8. doi: 10.1161/01.cir.97.5.425. PMID 9490235
- [Background] Criqui MH, Ho LA, Denenberg JO, Ridker PM, Wassel CL, McDermott MM. Biomarkers in peripheral arterial disease patients and near- and longer-term mortality. J Vasc Surg. 2010 Jul;52(1):85-90. doi: 10.1016/j.jvs.2010.02.004. Epub 2010 May 14. PMID 20471776
- [Background] Carriere I, Dupuy AM, Lacroux A, Cristol JP, Delcourt C; Pathologies Oculaires Liees a l'Age Study Group. Biomarkers of inflammation and malnutrition associated with early death in healthy elderly people. J Am Geriatr Soc. 2008 May;56(5):840-6. doi: 10.1111/j.1532-5415.2008.01677.x. Epub 2008 Apr 9. PMID 18410327
- [Background] Vidula H, Tian L, Liu K, Criqui MH, Ferrucci L, Pearce WH, Greenland P, Green D, Tan J, Garside DB, Guralnik J, Ridker PM, Rifai N, McDermott MM. Biomarkers of inflammation and thrombosis as predictors of near-term mortality in patients with peripheral arterial disease: a cohort study. Ann Intern Med. 2008 Jan 15;148(2):85-93. doi: 10.7326/0003-4819-148-2-200801150-00003. PMID 18195333
- [Background] Owens CD, Ridker PM, Belkin M, Hamdan AD, Pomposelli F, Logerfo F, Creager MA, Conte MS. Elevated C-reactive protein levels are associated with postoperative events in patients undergoing lower extremity vein bypass surgery. J Vasc Surg. 2007 Jan;45(1):2-9; discussion 9. doi: 10.1016/j.jvs.2006.08.048. Epub 2006 Nov 21. PMID 17123769
- [Background] Conen D, Rexrode KM, Creager MA, Ridker PM, Pradhan AD. Metabolic syndrome, inflammation, and risk of symptomatic peripheral artery disease in women: a prospective study. Circulation. 2009 Sep 22;120(12):1041-7. doi: 10.1161/CIRCULATIONAHA.109.863092. Epub 2009 Sep 8. PMID 19738135
- [Background] Havelka GE, Kibbe MR. The vascular adventitia: its role in the arterial injury response. Vasc Endovascular Surg. 2011 Jul;45(5):381-90. doi: 10.1177/1538574411407698. Epub 2011 May 13. PMID 21571779
- [Background] Inoue T, Croce K, Morooka T, Sakuma M, Node K, Simon DI. Vascular inflammation and repair: implications for re-endothelialization, restenosis, and stent thrombosis. JACC Cardiovasc Interv. 2011 Oct;4(10):1057-66. doi: 10.1016/j.jcin.2011.05.025. PMID 22017929
- [Background] Schillinger M, Exner M, Mlekusch W, Rumpold H, Ahmadi R, Sabeti S, Haumer M, Wagner O, Minar E. Vascular inflammation and percutaneous transluminal angioplasty of the femoropopliteal artery: association with restenosis. Radiology. 2002 Oct;225(1):21-6. doi: 10.1148/radiol.2251011809. PMID 12354979
- [Background] Brevetti G, Silvestro A, Di Giacomo S, Bucur R, Di Donato A, Schiano V, Scopacasa F. Endothelial dysfunction in peripheral arterial disease is related to increase in plasma markers of inflammation and severity of peripheral circulatory impairment but not to classic risk factors and atherosclerotic burden. J Vasc Surg. 2003 Aug;38(2):374-9. doi: 10.1016/s0741-5214(03)00124-1. PMID 12891123
- [Background] Busti C, Falcinelli E, Momi S, Gresele P. Matrix metalloproteinases and peripheral arterial disease. Intern Emerg Med. 2010 Feb;5(1):13-25. doi: 10.1007/s11739-009-0283-y. Epub 2009 Jul 21. PMID 19626421
- [Background] Owens CD, Wake N, Conte MS, Gerhard-Herman M, Beckman JA. In vivo human lower extremity saphenous vein bypass grafts manifest flow mediated vasodilation. J Vasc Surg. 2009 Nov;50(5):1063-70. doi: 10.1016/j.jvs.2009.06.022. Epub 2009 Aug 12. PMID 19679424
- [Background] Grenon SM, Conte MS, Nosova E, Alley H, Chong K, Harris WS, Vittinghoff E, Owens CD. Association between n-3 polyunsaturated fatty acid content of red blood cells and inflammatory biomarkers in patients with peripheral artery disease. J Vasc Surg. 2013 Nov;58(5):1283-90. doi: 10.1016/j.jvs.2013.05.024. Epub 2013 Jul 2. PMID 23830313
- [Background] Ho KJ, Spite M, Owens CD, Lancero H, Kroemer AH, Pande R, Creager MA, Serhan CN, Conte MS. Aspirin-triggered lipoxin and resolvin E1 modulate vascular smooth muscle phenotype and correlate with peripheral atherosclerosis. Am J Pathol. 2010 Oct;177(4):2116-23. doi: 10.2353/ajpath.2010.091082. Epub 2010 Aug 13. PMID 20709806
- [Background] Goodney PP, Beck AW, Nagle J, Welch HG, Zwolak RM. National trends in lower extremity bypass surgery, endovascular interventions, and major amputations. J Vasc Surg. 2009 Jul;50(1):54-60. doi: 10.1016/j.jvs.2009.01.035. Epub 2009 May 28. PMID 19481407
- [Background] Mahoney EM, Wang K, Keo HH, Duval S, Smolderen KG, Cohen DJ, Steg G, Bhatt DL, Hirsch AT; Reduction of Atherothrombosis for Continued Health (REACH) Registry Investigators. Vascular hospitalization rates and costs in patients with peripheral artery disease in the United States. Circ Cardiovasc Qual Outcomes. 2010 Nov;3(6):642-51. doi: 10.1161/CIRCOUTCOMES.109.930735. Epub 2010 Oct 12. PMID 20940249
- [Background] Sachs T, Pomposelli F, Hamdan A, Wyers M, Schermerhorn M. Trends in the national outcomes and costs for claudication and limb threatening ischemia: angioplasty vs bypass graft. J Vasc Surg. 2011 Oct;54(4):1021-1031.e1. doi: 10.1016/j.jvs.2011.03.281. Epub 2011 Aug 31. PMID 21880457
- [Background] Pande RL, Perlstein TS, Beckman JA, Creager MA. Secondary prevention and mortality in peripheral artery disease: National Health and Nutrition Examination Study, 1999 to 2004. Circulation. 2011 Jul 5;124(1):17-23. doi: 10.1161/CIRCULATIONAHA.110.003954. Epub 2011 Jun 20. PMID 21690489
- [Derived] Schaller MS, Chen M, Colas RA, Sorrentino TA, Lazar AA, Grenon SM, Dalli J, Conte MS. Treatment With a Marine Oil Supplement Alters Lipid Mediators and Leukocyte Phenotype in Healthy Patients and Those With Peripheral Artery Disease. J Am Heart Assoc. 2020 Aug 4;9(15):e016113. doi: 10.1161/JAHA.120.016113. Epub 2020 Jul 22. PMID 32696697